CLINICAL TRIAL: NCT05635721
Title: Influence of Different Ankle Positions on Nerve Conduction Parameters of Deep Peroneal Nerve
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Salah Abd-Elfattah, Demonstrator, Cairo University
Other Study IDs: P.T.REC/012/004076
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND:

The deep peroneal nerve arises as a branch of the common peroneal nerve which courses around the neck of the fibula. The motor component of deep peroneal nerve is responsible for innervating the anterior compartment of the lower leg which includes the tibialis anterior, extensor hallucis longus, extensor digitorum longus, and peroneus tertius muscles.

Nerve conduction velocity shortly known as "NCV" tests are used determine the speed of the electrical signals moving along a specific peripheral nerve .This will be helpful in localizing the site of entrapment of peripheral nerves and useful for assessing both recovery and prognosis of any injury to peripheral nervesthere are numerous aspects that could influence nerve conduction study.

Although changes in joint position have been reported in several studies to affect nerve conduction velocity of peripheral nerves. the effect of changing ankle joint position on deep peroneal NCV has not been repor Purpose

This study will investigate the effect of different ankle positions on:

1. Deep peroneal nerve distal motor latency across ankle joint.
2. Deep peroneal nerve sensory onset latency across ankle joint

DETAILED DESCRIPTION:
31healthy subjects of both genders with age ranging from 20to 40years old were examined for motor distal latency and sensory onset latency at three different ankle positions :neutral,20degrees dorsiflexion and 40degrees plantar flexion

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects.
* Age ranges from 20 to 40 years because longer latencies and slower nerve conduction velocity are seen significantly with increasing age.
* All participants will be selected with body mass index (BMI) between 18.5 and 24.9kg/cm2 .

Exclusion criteria:

* Elderly subjects.
* Pregnant women.
* Subjects with history of or risk factors for peripheral nerve lesions.
* Obese subjects.
* Subjects with any foot deformity.
* History of lower limb fractures.
* History of surgery to lower limbs
* Diabetic patients.
* Patients with cardiovascular disorders.
* Hypertensive patients.
* Women wearing high heeled shoes.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 31 healthy subjects of both genders will be recruited to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Deep peroneal nerve motor distal latency | 30 minutes for each participant
  Motor distal latency: It is the time between the distal stimulus and the onset of compound muscle action potential(CMAP)at recording muscles
Deep peroneal nerve sensory onset latency | 30 minutes for each participant
  : It is the time taken from the stimulus artifact to the initial negative deflection of the sensory nerve action potential (SNAP)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Salah, Principal Investigator — faculty of physical therapy
Locations (1):
- Mahmoud Salah, Aga, Egypt